CLINICAL TRIAL: NCT03321955
Title: Prospective Study of Conservative Ziconotide Dosing as a First-Line Intrathecal Drug Therapy for Neuropathic Pain
Brief Title: Ziconotide as First-Line IDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Julie Pilitsis, MD, MD, Albany Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jazz Prospective
Record Dates: First submitted 2017-10-19; First posted 2017-10-26 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — ziconotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Subjects with Painful Neuropathy (Experimental): All subjects will be implanted with the Medtronic Synchromed II pump, and treated with the same algorithm for dose adjustment for painful neuropathy with Ziconotide 100 micrograms/ml.
  Interventions: Drug: Ziconotide 100 MCG(microgram)/ML Intrathecal Solution; Diagnostic Test: Quantitative sensory testing; Diagnostic Test: Serum markers: Interleukin-1, Interleukin-6, and tumor necrosis factor

INTERVENTIONS:
Drug: Ziconotide 100 MCG(microgram)/ML Intrathecal Solution — Initial dose at time of the implant will be 1.2 mcg/day with dose increases of no more the .4 mcg/day planned for 3, 6, 8, 9, 10, 12 weeks and 4, 5, 6 and 12 months.
Diagnostic Test: Quantitative sensory testing — Quantitative sensory testing will be done using different types of sensory stimulation to objectively quantify sensation and pain tolerance. VonFrey fibers of various widths are used to detect sensation, a Neuropen pin prick iutilized to detect pain, along with a tuning fork to measure vibrationand a pressure guage to measure pressure felt on the skin. Cold/hot sensation is tested with Medoc Pathway system to quantitatively measure the temperature felt by patients to be done at baseline, 6 months and 12 months,
Diagnostic Test: Serum markers: Interleukin-1, Interleukin-6, and tumor necrosis factor — Increases in these biomarkers indicate nerve pain as they are released from macrophages in patients with damaged nerves.

SUMMARY:
The primary objective of this study is to prospectively examine outcomes in 12 patients using ziconotide Intrathecal Drug Therapy(IDT) as first-line monotherapy with the use of an algorithm of slow titration for dosing. The use of Prialt has demonstrated fewer and less serious associated adverse effects as compared to IDT morphine, especially when titrated slowly. We will use an average Numerical Rating Scale as our primary outcome and the Oswestry Disability Index(ODI), Beck Depression Inventory (BDI), Pain Catastrophizing Scale (PCS), Clinical Global Impression of Change Scale including binary satisfaction measures(CGIC), Lawton-Brody Instrumental Activities of Daily Living(IADL) and Short Form-36 as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Must be eligible for implantation of an intrathecal analgesia programmable pump system using ziconotide IT.
2. Must be 18 years of age or older for all points of data collection.
3. Must be diagnosed with neuropathic pain secondary to a clear etiology. Acceptable etiologies including but not limited to diabetic neuropathy, small fiber neuropathy, and post herpetic neuropathy.

Exclusion Criteria:

1. Must not have or been previously implanted with a programmable pump system.
2. Untreated mental illness including depression or anxiety determined by preoperative psychological evaluation.
3. Active substance abuse determined by preoperative urine drug screen.
4. Unwillingness to decrease oral medications at screening.
5. Any prior use of intrathecal analgesia besides trialing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | Baseline, 3, 4, 6, 8, 9, 10, 12 week and 4, 5, 6 and 12 months
  This scale allows the subject to quantify their pain numerically, with 10 being the worst pain imaginable. This scale describe subject reported pain at its worst and best in the week prior to reporting, as well as total pain on average, and at the time of documentation. The mean of these scores will be used as the primary outcome. This scale also includes a question of subject experienced global improvement in which the patient is asked to quantify their overall change in pain with 0 being no change and 10 being completely changed. Using the NRS we will calculate a responder rate, assessing percentage of patients with a 50% response in NRS

SECONDARY OUTCOMES:
Oswestry Disability Index Scale | Baseline, 12 weeks, 6 month, 12 month
  Comprises 11 sections, this survey asks the patient to indicate the degree to which they have difficulty in daily life relating to pain.
SF (Short Form) - 36 | Baseline, 12 weeks, 6 month
  This scale utilizes 36 questions to determine overall quality of life in patients by discussing physical health, emotional health, and social engagement.
IADL(Instrumental Activities of Daily Living) | Baseline, 12 weeks, 6 month, 12 month
  Used to assess complex functional activities of daily living, this scale extrapolates on basic activities such as ability to eat or walk, to include cooking shopping, housekeeping.
Beck Depression Inventory | Baseline, 12 weeks, 6 month, 12 month
  21 question survey pertaining to a patient's severity of depression. Each question is scored for 0 to 3, with 0 indicating no depression and 3 indicating the most severe depression
Pain Catastrophizing Scale | Baseline, 12 weeks, 6 month, 12 month
  This scale separates three types of catastrophizing: rumination, magnification and helplessness. Catastrophic thinking can contribute to the probability that a pain condition will be persistent over tim.

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College, Albany, New York, United States